CLINICAL TRIAL: NCT05587140
Title: Effects of Conventional Versus Acupuncture-like TENS on Pain Threshold and Brain Activities in Healthy Adults
Brief Title: Effects of TENS on Pain Threshold and Brain Activities in Healthy Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: TENS & pain control
Record Dates: First submitted 2022-07-10; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-06

CONDITIONS: Transcutaneous Electrical Nerve Stimulation; Electroencephalography; Pressure Pain Threshold
Keywords: Transcutaneous electrical nerve stimulation; Electroencephalography; Pressure pain threshold; Pressure pain tolerance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupuncture like TENS (Experimental): The study would use acupuncture like TENS for 30 minutes
  Interventions: Device: Acupuncture like TENS
- Conventional TENS (Experimental): The study would use conventional TENS for 30 minutes
  Interventions: Device: Conventional TENS
- Sham TENS (Experimental): The study would use sham TENS for 30 minutes
  Interventions: Device: Sham TENS

INTERVENTIONS:
Device: Acupuncture like TENS — Frequency: 4 Hz, pulse duration: 200 μs, intensity: 3/10 painful sensation with muscle contraction , time: 30 minutes
  Arms: Acupuncture like TENS
Device: Conventional TENS — Frequency: 100 Hz, pulse duration: 200 μs, intensity: strong but comfortable tingling sensation , time: 30 minutes
  Arms: Conventional TENS
Device: Sham TENS — Frequency: 4 Hz, pulse duration: 200 μs, intensity: tingling sensation, time: turn on the electricity for 15 seconds, then turn off the machine for 30 minutes
  Arms: Sham TENS

SUMMARY:
The purpose of this study was to understand the effects of conventional versus acupuncture-like TENS on pain threshold, brain activities, and their relationships.

DETAILED DESCRIPTION:
Transcutaneous electrical nerve stimulation (TENS) is a pain modulation tool which is commonly used clinically. TENS has 2 major modes: "conventional TENS'' and "acupuncture like TENS". Conventional TENS induces a local pain modulation, whereas acupuncture like TENS induces central pain modulation mechanism. The pain threshold at treatment area and outside of area is regarded as local pain modulation and central pain modulation respectively. However, the effect of acupuncture like TENS on pain threshold was remained unclear. TENS also induces cortical activities changed in the central nervous system. Recent Electroencephalography (EEG) studies suggested that TENS induces event-related potential and power spectrum changes, however, the time and frequency bands of EEG changes and its relationship with pain threshold were still unclear. Therefore, the purpose of this study was to understand the effects of conventional versus acupuncture-like TENS on pain threshold, brain activities, and their relationships.

ELIGIBILITY:
Inclusion Criteria:

* 20~65 y adults
* No cognitive function problem
* Without taking any type of pain medication or substances that could affect the cognitive functions

Exclusion Criteria:

* Peripheral or central nervous system disease
* Sensory lose
* TENS application is contraindication
* Cardiac pacemaker
* Any type of pain

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Pressure pain threshold after the intervention | The change between baseline and the time after 30 minutes intervention
  Use a pressure algometer to press on the first dorsal interosseous muscle and the pressure would stop until the feeling changes from non-painful feeling to painful feeling.
Pressure pain tolerance after the intervention | The change between baseline and the time after 30 minutes intervention
  Use a pressure algometer to press on the first dorsal interosseous muscle and the pressure would stop until the feeling reach the pain intensity at 5/10.
EEG power spectrum change in delta band after the intervention | The change between baseline and the time after 30 minutes intervention
  Evaluate brain activity after the intervention
EEG power spectrum change in theta band after the intervention | The change between baseline and the time after 30 minutes intervention
  Evaluate brain activity after the intervention
EEG power spectrum change in alpha band after the intervention | The change between baseline and the time after 30 minutes intervention
  Evaluate brain activity after the intervention
EEG power spectrum change in beta band after the intervention | The change between baseline and the time after 30 minutes intervention
  Evaluate brain activity after the intervention
EEG power spectrum change in low-gamma band after the intervention | The change between baseline and the time after 30 minutes intervention
  Evaluate brain activity after the intervention
EEG power spectrum change in high-gamma band after the intervention | The change between baseline and the time after 30 minutes intervention
  Evaluate brain activity after the intervention
EEG power spectrum change in total gamma band after the intervention | The change between baseline and the time after 30 minutes intervention
  Evaluate brain activity after the intervention

SECONDARY OUTCOMES:
Pressure pain tolerance after the 30 minutes break | The change between 30 minutes intervention and 30 minutes break after the intervention
  Use a pressure algometer to press on the first dorsal interosseous muscle and the pressure would stop until the feeling reach the pain intensity at 5/10.
Pressure pain threshold after the 30 minutes break | The change between 30 minutes intervention and 30 minutes break after the intervention
  Use a pressure algometer to press on the first dorsal interosseous muscle and the pressure would stop until the feeling changes from non-painful feeling to painful feeling.
EEG power spectrum change in delta band after the 30 minutes break | The change between 30 minutes intervention and 30 minutes break after the intervention
  Evaluate brain activity after the 30 minutes break
EEG power spectrum change in theta band after the 30 minutes break | The change between 30 minutes intervention and 30 minutes break after the intervention
  Evaluate brain activity after the 30 minutes break
EEG power spectrum change in alpha band after the 30 minutes break | The change between 30 minutes intervention and 30 minutes break after the intervention
  Evaluate brain activity after the 30 minutes break
EEG power spectrum change in beta band after the 30 minutes break | The change between 30 minutes intervention and 30 minutes break after the intervention
  Evaluate brain activity after the 30 minutes break
EEG power spectrum change in low-gamma band after the 30 minutes break | The change between 30 minutes intervention and 30 minutes break after the intervention
  Evaluate brain activity after the 30 minutes break
EEG power spectrum change in high-gamma band after the 30 minutes break | The change between 30 minutes intervention and 30 minutes break after the intervention
  Evaluate brain activity after the 30 minutes break
EEG power spectrum change in total gamma band after the 30 minutes break | The change between 30 minutes intervention and 30 minutes break after the intervention
  Evaluate brain activity after the 30 minutes break

CONTACTS AND LOCATIONS:
Overall Officials: Li-Wei Chou, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang-Ming University, Taipei, Taiwan